CLINICAL TRIAL: NCT03010020
Title: STI Screening as a Combined HIV Prevention Platform for MSM in Peru
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: NGO Via Libre (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Jesse Clark, Associate Professor-in-Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R34MH105272 (NIH)
Record Dates: First submitted 2017-01-01; First posted 2017-01-04 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Gonorrhoea of Rectum; Chlamydia of Rectum; HIV Infections
Keywords: HIV Prevention; MSM; Rectal Gonorrhea; Rectal Chlamydia; Personalized Cognitive Counseling
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STI-Positive: PCC (Experimental): MSM diagnosed with rectal GC and/or CT infection counseled for HIV prevention using Personalized Cognitive Counseling (PCC) and treated with appropriate antibiotic therapy
  Interventions: Behavioral: PCC
- STI-Positive: Traditional Counseling (Placebo Comparator): MSM diagnosed with rectal GC and/or CT infection counseled for HIV prevention using traditional risk reduction counseling and treated with appropriate antibiotic therapy
  Interventions: Behavioral: Traditional Counseling
- STI-Negative (No Intervention): MSM without rectal GC and/or CT infection

INTERVENTIONS:
Behavioral: PCC — Personalized Cognitive Counseling (PCC) sessions will be delivered as described above.
  Arms: STI-Positive: PCC
Behavioral: Traditional Counseling — GC/CT-infected participants in the standard of care arm (and all GC/CT-negative participants screened for infection) will receive standard post-test counseling in accordance with Peruvian Ministry of Health guidelines.
  Arms: STI-Positive: Traditional Counseling

SUMMARY:
The investigators propose to develop and pilot an HIV prevention intervention based on rectal STI testing, counseling, and treatment for MSM in Peru. The investigators will use nucleic acid testing to screen 750 behaviorally high-risk MSM for rectal gonorrheal and/or chlamydial (GC/CT) infection. GC/CT-positive subjects will receive single-dose antibiotic treatment and single-session Personal Cognitive Counseling (PCC) (n=50) or standard post-test counseling (n=50). A GC/CT-negative control group (n=50) will also be enrolled to compare biological outcomes including changes in levels of inflammatory cytokines following rectal STI. The intervention is based on three interrelated objectives: 1) To use periodic rectal STI nucleic acid testing to identify the members of the MSM population at greatest short-term risk for HIV infection; 2) To provide single-dose antibiotic treatment to control the immune activation and mucosal inflammation caused by rectal GC/CT infection that increase cellular risk for HIV transmission; and 3) To use Personal Cognitive Counseling (PCC) to understand and modify recent high-risk sexual practices that led to rectal STI acquisition and that increase future HIV risk.

The investigators propose to screen 750 behaviorally high-risk MSM for rectal GC/CT infection to enroll 100 GC/CT-positive individuals (using a conservative 15% prevalence estimate) and 50 GC/CT-negative controls (matched by age and baseline frequency of URAI). GC/CT-infected participants will be given single-dose antibiotic therapy and randomized to receive single-session PCC (n=50) or standard post-test counseling (n=50). The primary outcome will be the impact of PCC on self-reported sexual risk behavior (URAI). Secondary outcomes will assess: 1) Feasibility/Acceptability of the STI screening program; 2) Impact of GC/CT infection and treatment on levels of inflammatory cytokines (IL-6, IL-8, TNF-αand IL-1β) in rectal mucosa; 3) Prevalence of persistent/recurrent rectal GC/CT; and 4) HIV incidence in GC/CT-infected and -uninfected MSM.

DETAILED DESCRIPTION:
Overview. The investigators plan to screen 750 behaviorally high-risk, HIV-uninfected MSM in order to enroll 100 subjects with rectal GC/CT infection and 50 uninfected controls. GC/CT-infected participants will receive single-dose antibiotic therapy and be randomized to receive either PCC or standard-of-care post-test counseling. GC/CT-negative participants will receive standard post-test counseling. Behavioral and biological assessments will be conducted at Baseline, 3-month and 6-month Follow-up visits. The primary outcome will be the effect of PCC on the prevalence of URAI with an HIV-infected or unknown status partner in the preceding 3-months. Secondary outcomes include feasibility/acceptability of the intervention, prevalence of persistent or recurrent GC/CT infection, change in rectal cytokine levels, and incidence of HIV infection.

Recruitment. Participants will be recruited from local HIV testing sites using the methods described above.

Screening Visit. The investigators will screen 750 MSM reporting at least one recent episode of unprotected receptive anal intercourse (URAI) for rectal GC/CT infection with a goal of identifying 100 GC/CT-positive participants (using a conservative 15% prevalence estimate and assuming 10% loss to follow-up over 6 months).

i) Rapid HIV Testing: After providing informed consent, all potential participants will undergo rapid HIV testing. Study staff will provide pre- and post-test risk reduction counseling based on the CDC's RESPECT-2 model (24) and screen for HIV at point of care using a 4th Generation Rapid HIV-1/2 assay (Alere Determine, Alere).

ii) Physical Examination: Potential participants will undergo routine physical examination to assess for signs of STI. Participants with evidence of proctitis (rectal discharge or inflammation) will be treated with Ceftriaxone 250 mg injection and Azithromycin 1 g oral and invited to enroll in the study based on symptomatic criteria.

iii) Syphilis Testing: Potential participants will undergo syphilis testing by RPR (RPRnosticon, Biomerieux), with positive results confirmed by TPPA (Serodia TPPA, Fujirebio). Results will be provided within 14 days and individuals with latent syphilis infection will be treated with three weekly doses of Penicillin G 2.4 Million IU.

iv) Rectal NAT Screening: All potential participants, regardless of symptoms, will be tested for rectal GC/CT infection at the screening visit. A rectal swab will be obtained by clinical staff and tested for GC/CT using a transcription mediated assay (TMA) (GenProbe Aptima, Hologic). Results will be provided within 14 days.

v) Antibiotic Therapy: Participants with symptomatic proctitis at the screening visit will be provided with appropriate antibiotic treatment (Ceftriaxone 250 mg IM and Azithromycin 1g PO once), advised of the importance of partner notification, and offered antibiotic therapy packets to deliver to their recent sexual partners (maximum of 5 packets per participant). Each packet will include a single dose of Cefixime 400 mg and Azithromycin 1g PO as well as printed information about GC/CT infection and local testing and treatment resources for HIV and other STIs (including free partner testing and treatment at the Via Libre site).

Enrollment Visit. Based on results of nucleic acid testing and/or symptomatic criteria, we will enroll 100 HIV-uninfected MSM with rectal GC/CT infection who will be randomized to receive either PCC (n=50) or standard post-test counseling (n=50). An additional 50 GC/CT-uninfected control subjects will also be enrolled.

i) Antibiotic Therapy: Participants diagnosed with rectal GC/CT by nucleic acid testing will receive antibiotic therapy and up to 5 partner treatment packets as described above.

ii) Randomization: Participants diagnosed with rectal GC/CT infection and/or symptomatic proctitis will be randomized to receive either PCC or standard of care post-test counseling. Randomization assignments will be constructed in a random permuted block allocation (block size = 7, alternating 4/3 ratio). Computer-generated assignments will be stored in opaque, sealed envelopes and opened sequentially at the time of allocation.

iii) Behavioral Survey: GC/CT-infected participants in both arms will be asked to complete a CASI-administered behavioral survey. The survey instrument will be self-administered using an iPad device and will ask participants about their sexual practices during the previous 3 months, including number and type of sexual partners (primary/stable partner, casual/recurrent contact, casual/single contact, anonymous contact, and commercial sex client or worker), frequency of sexual intercourse (oral, anal, and vaginal), frequency of unprotected intercourse, and frequency of unprotected intercourse with HIV-infected or unknown serostatus partners. To collect additional detail on partner-level risk factors, participants will be asked to provide information about their most recent sexual contacts (up to a maximum of three contacts within 6 months). For each contact, participants will be asked to describe the partner's age, gender, sexual orientation, sexual role, partnership type, length of partnership, partner HIV serostatus, and sexual practices, including act-specific condom use. Additional questions will address demographics, STI symptoms (e.g., dysuria, urethral or rectal discharge, etc.), drug and alcohol use, depression, anxiety, and self-efficacy for negotiating condom use.

iv) Personal Cognitive Counseling (PCC): After completing the survey, participants diagnosed with GC/CT-infection will receive either PCC or standard of care post-test counseling, according to randomization arm.

PCC Procedures: i) SJEI Completion: Participants will first be asked to complete the SJEI instrument independently. ii) SJEI Review: A study counselor will meet with the participant to review their responses to the SJEI and ask them to recount a recent sexual encounter involving URAI. Participants will be asked to tell their story in context, paying attention to the environmental cues, interpersonal interactions, and individual emotions and cognitive processes occurring at each step of the encounter. After narrating their story, the participant will review together with the counselor the self-justifications employed during the interaction, using objective, "offline" analysis to explore the "online" cognitive processes they used to justify sexual risk behavior during the episode. iii) Risk Counseling: The counselor will work with the participant to highlight moments where critical behavioral decision points occurred, identify the self-justifications used for engaging in risk behavior at those moments, and develop a strategy to control risk behavior in future interactions. A key component of the counseling will involve linking the prior episode of URAI with the current diagnosis of rectal GC/CT, as a strategy to highlight flaws in previously used self-justifications. iv) Role-Play: The counselor and the participant will rehearse risk reduction strategies by role-playing typical interactions where high-risk sexual behavior may occur. After completing the session, the participant will be asked to discuss their satisfaction with the PCC model, including their comfort in discussing the cognitive processes occurring during a sexual encounter, the perceived usefulness of the counseling, and any important issues that were not addressed.

v) Standard of Care Post-Test Counseling. GC/CT-infected participants in the standard of care arm (and all GC/CT-negative participants screened for infection) will receive standard post-test counseling in accordance with Peruvian Ministry of Health guidelines. Counseling will include a discussion of recent sexual risk behavior, condom use to reduce the risk of future HIV/STI acquisition, partner notification, and follow-up testing.

vi) Rectal Cytokine Measurements. GC/CT-infected participants randomized to the standard post-test counseling arm will be matched 1-to-1 with GC/CT-negative controls. Matching will be based on age and number of episodes of URAI reported in the previous 30 days (categorized as 1, 2-3, or >3 episodes).

GC/CT-infected participants and matched GC/CT-negative controls will be asked to provide a swab sample of the rectal mucosa to monitor changes in levels of inflammatory cytokines from the time of diagnosis to after antibiotic treatment. To collect the sample, a physician will insert a sponge swab 4 cm into the participant's rectum and leave it in place for 30 seconds prior to removal. Samples will be stored in liquid transport media at -4°C until completion of the study, at which time all samples will be sent to the UCLA Mucosal Immunology Core (MIC) Laboratory. Levels of IL-1β, IL-6, IL-8, and TNF-α in rectal mucosa will be measured. Repeat measurements will be collected at 3- and 6-month Follow-up visits to assess changes from initial diagnosis to post-treatment. Results will be used to establish baseline values and changes in levels of key cytokines following STI treatment to define the parameters for intermediate biological outcomes in a projected RCT.

Follow-up Visits. All participants will be asked to return for 3-month and 6-month Follow-up assessments.

i) Behavioral Survey. All participants diagnosed with rectal GC/CT infection at Enrollment will be asked to complete a CASI-administered Follow-up survey at each visit. Similar to the Baseline survey, the Follow-up instrument will assess sexual risk behavior, substance use, and other mediating factors (depression, anxiety, condom self-efficacy) over the previous 3-month period as well as partner notification and treatment outcomes.

ii) Repeat HIV Testing. Rapid HIV testing will be provided at each follow-up visit using the above procedures.

iii) Repeat GC/CT Testing. All participants will receive repeat nucleic acid testing for rectal GC/CT at each follow-up visit. Results of repeat testing will be provided by telephone or in person within two weeks. Participants with new, recurrent, or persistent infection will be treated with Ceftriaxone 250 mg IM and Azithromycin 1g PO once. Post-test counseling for new, persistent, or recurrent infection will be provided according to the participant's original randomization assignment (PCC or standard of care counseling).

iv) Repeat Cytokine Testing. Rectal swab measurements will be obtained from GC/CT-positive participants randomized to the standard of care arm and matched GC/CT-negative controls at each follow-up to monitor changes in inflammatory cytokine levels in rectal mucosa after antibiotic treatment and in GC/CT-negative controls over the same time period. Samples will be stored for testing in the UCLA MIC laboratory.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Assigned male sex at birth
* HIV-uninfected
* Reports receptive anal intercourse with an HIV-infected or unknown serostatus partner within the previous 6 months
* Diagnosed with rectal gonorrhea and/or chlamydia infection (not applicable to GC/CT-uninfected controls)

Exclusion Criteria:

* Unable to complete informed consent procedures
* HIV-infected (according to laboratory testing)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Unprotected Receptive Anal Intercourse (URAI) with Serodiscordant or Unknown Serostatus Partner | 6 Months
  prevalence of self-reported URAI with an HIV-infected or unknown serostatus partner at 6-month Follow-up

SECONDARY OUTCOMES:
Persistent or Recurrent Rectal GC/CT Infection | 6 Months
  Effect of the intervention on the prevalence of persistent or recurrent rectal GC/CT infection will be assessed through repeat nucleic acid testing at 3- and 6-month Follow-up.
Inflammatory Cytokine Levels in Rectal Mucosa | 6 Months
  Levels of IL-1β, IL-6, IL-8, and TNF-α in rectal mucosa will also be measured at Enrollment and 3- and 6-month Follow-up. Average levels of inflammatory cytokines in individuals with rectal GC/CT infection will be measured at time of diagnosis and after antibiotic treatment, and compared with GC/CT-negative controls.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse L Clark, MD, MSc, Principal Investigator — University of California, Los Angeles
Locations (1):
- Asociacion Civil Via Libre, Lima, Peru

IPD SHARING:
Plan to Share IPD: No
Due to restrictions on access to human subjects data, data will be made available to other researchers upon request and approval by the governing IRB/Ethics Committee.

REFERENCES:
- [Derived] Clark JL, Oldenburg CE, Passaro RC, Segura ER, Godwin W, Fulcher JA, Cabello R. Changes in Inflammatory Cytokine Levels in Rectal Mucosa Associated With Neisseria gonorrheae and/or Chlamydia trachomatis Infection and Treatment Among Men Who Have Sex With Men in Lima, Peru. J Infect Dis. 2024 Mar 14;229(3):845-854. doi: 10.1093/infdis/jiad349. PMID 37584273
- [Derived] Ayer A, Segura ER, Perez-Brumer A, Chavez-Gomez S, Fernandez R, Gutierrez J, Suarez K, Lake JE, Clark JL, Cabello R. Sexual health norms and communication patterns within the close social networks of men who have sex with men and transgender women in Lima, Peru: a 2017 cross-sectional study. BMC Public Health. 2021 Jun 7;21(1):1090. doi: 10.1186/s12889-021-11091-2. PMID 34098916
- [Derived] Blair CS, Lake JE, Passaro RC, Chavez-Gomez S, Segura ER, Elliott J, Fulcher JA, Shoptaw S, Cabello R, Clark JL. Brief Report: HIV-1 Seroconversion Is Not Associated With Prolonged Rectal Mucosal Inflammation. J Acquir Immune Defic Syndr. 2021 Apr 15;86(5):e134-e138. doi: 10.1097/QAI.0000000000002601. PMID 33351532
- [Derived] Passaro RC, Castaneda-Huaripata A, Gonzales-Saavedra W, Chavez-Gomez S, Segura ER, Lake JE, Cabello R, Clark JL. Contextualizing condoms: a cross-sectional study mapping intersections of locations of sexual contact, partner type, and substance use as contexts for sexual risk behavior among MSM in Peru. BMC Infect Dis. 2019 Nov 11;19(1):958. doi: 10.1186/s12879-019-4517-y. PMID 31711433